CLINICAL TRIAL: NCT07168564
Title: Post Market Clinical Study to Compare Vision With Essilor® AVA™ Lenses Following AVA™ Refraction Protocol to Equivalent Lenses Following Gold Standard Refraction Protocol.
Brief Title: Post Marketing Clinical Study on the Efficacy of Lenses From a New Prescription Protocol
Acronym: ATLANTIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Essilor International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: WS10425
Record Dates: First submitted 2025-08-26; First posted 2025-09-11 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-10

CONDITIONS: Ametropia; Refractive Error
Keywords: Corrective eye glasses
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Intervention Model Description: Post-Marketing Clinical Study : Monocentric, 2 arms, crossover, prospective, interventional, double masked clinical study, with within-subject control
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- First Essilor® AVA™ and then Standard (Experimental): Participants are first prescribed for AVA™ protocol and then for Standard protocol . Patients will first wear the Essilor® AVA™ lenses during 2 weeks. Then, after a washout period of 2 weeks, patients will wear the Standard lenses during 2 weeks.
  Interventions: Device: AVA lenses; Device: Standard lenses
- First Standard then Essilor® AVA™ (Experimental): Participants are first prescribed for Standard protocol and then for AVA™ protocol . Patients will first wear the Standard lenses during 2 weeks. Then, after a washout period of 2 weeks, patients will wear the Essilor® AVA™ lenses during 2 weeks.
  Interventions: Device: AVA lenses; Device: Standard lenses

INTERVENTIONS:
Device: AVA lenses — Participants are prescribed to receive AVA lenses through the AVA protocol and wear these lenses during 2 weeks.
Device: Standard lenses — Participants are prescribed to receive Standard lenses through the Gold standard protocol and wear these lenses during 2 weeks.

SUMMARY:
The goal of this clinical trial is to assess improvements in visual performance and patient outcomes in wearing new spectacle lenses in general population.

The two spectacle lenses will be compared after two weeks of wearing.

The aims are:

* to evaluate the visual superiority, and quality-of-life implications of Essilor® AVA™ spectacle lenses prescribed after a new subjective refraction protocol named AVA™ protocol.
* to understand the benefits of using a high accuracy instrument and testing sequence over the standard testing sequence in determining a glasses prescription, as well as the overall subjective performance of the resulting glasses.

DETAILED DESCRIPTION:
This study aims to evaluate whether finer increments in refraction and spectacle lens manufacturing (0.01D) provide more precise visual corrections compared to the traditional 0.25D steps, and if participants can visually appreciate this difference in the refractive outcome and manufactured lenses. It will assess improvements in visual acuity, comfort, and patient satisfaction, focusing on achieving red-green equality in the duo chrome test and exploring the clinical utility of higher resolution refraction technologies.

Refraction is a critical procedure in eye care that determines the optimal lens power for a focused retinal image. Traditional manual phoropters, the standard for over a century, operate in 0.25D increments but have limitations, as most individuals are sensitive to smaller power variations. Recent technological advancements, such as digital phoropters like the Vision-R™ 800, allow for continuous power adjustments in increments as fine as 0.01D and support manufacturing spectacles in smaller steps.

While these innovations offer theoretical advantages, their clinical impact remains relatively underexplored. This study addresses this gap by comparing traditional and finer increment prescriptions to assess improvements in visual performance and patient outcomes. Results could redefine refraction standards and optimize optometric care practices.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 y/o and 70
2. Accepted and signed the consent form
3. Agree to participate in the scheduled visits
4. Best-corrected visual acuity by manifest refraction of +0.10 log MAR (20/25 Snellen) or better in each eye
5. Spherical Equivalent Refractive Error between -10.00 and 10.00 D
6. Possess current wearable and visually functional eyeglasses
7. Agree to wear the assigned frames fitted with the provided lenses for a minimum of 14 days, during 6h/day, equivalent to 42 hours of wearing a week.
8. No binocular vision issues
9. No cataract, grade 2 or greater

   Presbyope subjects: To be eligible for the presbyopic group, individuals need to be (half of the analyzed population):
10. 35-70 years of age, inclusive
11. Currently wearing and adapted to progressive addition lenses

Exclusion Criteria:

1. Less than 18 years or greater than 70 years of age
2. Does not wear spectacles at least 6 hours/day
3. Does not have a wearable pair of glasses with a prescription ≤2 years old
4. Currently or formerly a licensed optometrist, optician, or ophthalmic technician trained in refraction

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-09-22 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Vision correction preference | through study completion, an average of 8 weeks
  Proportion of subjects preferring vision correction option between Essilor® AVA™ lenses and the alternative vision correction solution

SECONDARY OUTCOMES:
Subjective Binocular Vision Quality | immediately after the intervention, and through study completion, an average of 8 weeks
  Scores of self-reported Subjective Binocular Vision Quality questionnaire OU (0-100 rating) at Distance vision, Near work and Overall Quality of Vision.
Subjective Binocular Vision | immediately after the intervention, and through study completion, an average of 8 weeks
  P-value of superiority Wilcoxon signed rank test comparing the Scores regarding Subjective Binocular Vision obtained with Essilor® AVA™ lenses and with Essilor® non-AVA™ lenses
Accuracy of refraction | immediately after the intervention, and through study completion, an average of 8 weeks.
  Scores of self-reported perceived accuracy of refraction OU (0-100 rating) obtained with AVA™ Smart program and with standard refraction.
accuracy of refraction | immediately after the intervention, and through study completion, an average of 8 weeks.
  P-value of superiority Wilcoxon signed rank test comparing the Scores of self-reported perceived accuracy of refraction OU (0-100 rating) obtained with AVA™ Smart program and with standard refraction
perceived refraction experience | immediately after the intervention
  Score of self-reported perceived refraction experience of refraction OU (0-100 rating) obtained with AVA™ Smart program and with standard refraction.
Refraction experience accuracy of refraction | through study completion, an average of 8 weeks.
  P-value of superiority Wilcoxon signed rank test comparing the Scores of self-reported refraction experience accuracy of refraction OU (0-100 rating) obtained with AVA™ Smart program and with standard refraction.
Subjective refraction experience | immediately after intervention
  Score of self-reported Subjective refraction experience with Essilor® AVA™ lenses in following 2 weeks of wear - Comparison in High contrast, high illumination logMAR Visual Acuity (4m, OU (M&S)) with refractive outcome (superiority test)
Subjective Vision Quality with Essilor® AVA™ lenses | immediately after intervention, through study completion, an average of 8 weeks.
  P-value of superiority Wilcoxon signed rank test comparing the Scores of self-reported Subjective Vision Quality with Essilor® AVA™ lenses in following 2 weeks of wear - Comparison in High contrast, high illumination logMAR Visual Acuity (4m, OU (M&S)) with refractive outcome (superiority test)
Binocular high-contrast, high-illumination logMAR distance visual acuity | immediately after intervention, through completion of study, an average of 8 weeks.
  Binocular high-contrast, high-illumination logMAR distance visual acuity with AVA™ lenses and Vision-R™ 800.
binocular high-contrast high-illumination distance visual acuity | immediately after intervention, through completion of study, an average of 8 weeks.
  P-value of superiority Wilcoxon signed rank test comparing binocular high-contrast high-illumination distance visual acuity with the AVA™ Smart Program refraction results and Essilor® AVA™ lenses manufactured from this prescription, over the standard refraction results and corresponding Essilor® non-AVA™ lenses.
Binocular low-contrast high-illumination distance logMAR visual acuity | immediately after intervention, through completion of study, an average of 8 weeks.
  Binocular low-contrast high-illumination distance logMAR visual acuity with Essilor® AVA™ lenses and Vision-R 800™.
binocular low-contrast high-illumination distance log MAR visual acuity | immediately after intervention, through completion of study, an average of 8 weeks.
  P-value of superiority Wilcoxon signed rank test comparing binocular low-contrast high-illumination distance log MAR visual acuity with the AVA™ Smart Program refraction results and Essilor® AVA™ lenses manufactured from this prescription over the standard refraction results and corresponding Essilor® non-AVA™ lenses
Binocular low-contrast low-illumination distance logMAR visual acuity | immediately after intervention, through completion of study, an average of 8 weeks.
  Binocular low-contrast low-illumination distance logMAR visual acuity with Essilor® AVA™ lenses and Vision-R 800™.
binocular low-contrast low-illumination distance log MAR visual acuity | immediately after intervention, through completion of study, an average of 8 weeks.
  P-value of superiority Wilcoxon signed rank test comparing binocular low-contrast low-illumination distance log MAR visual acuity with the AVA™ Smart Program refraction results and Essilor® AVA™ lenses manufactured from this prescription over the standard refraction results and corresponding Essilor® non-AVA™ lenses.
Binocular distance contrast sensitivity | immediately after intervention, through completion of study, an average of 8 weeks.
  Binocular distance contrast sensitivity (4m, OU) with refractive outcome.
Binocular distance contrast sensitivity | immediately after intervention, through completion of study, an average of 8 weeks.
  P-value of superiority Wilcoxon signed rank test comparing Binocular distance contrast sensitivity with the AVA™ Smart Program refraction results and Essilor® AVA™ lenses manufactured from this prescription over the standard refraction results and Essilor® non-AVA™ lenses.
binocular stereo acuity | immediately after intervention
  Summarize binocular stereo acuity with AVA™ lenses and Vision-R 800™
binocular stereo acuity | immediately after intervention
  Mean difference in binocular stereo acuity (4m, Vision-R 800™ system) with the AVA™ Smart Program refraction results and prescribed Essilor® AVA™ lenses over the standard refraction results and corresponding Essilor® non-AVA™ lenses.
Duochrome Equality | immediately after intervention
  Summarize relative frequency of Duochrome Equality OD, OS in distance refractive outcomes
relative frequency of Duochrome Equality | through study completion, an average of 8 weeks.
  P-value of McNemar test comparing the relative frequency of Duochrome Equality OD, OS with AVA™ Smart Program refraction and with the standard refraction.
5-point Likert | through study completion, an average of 8 weeks.
  P-value of Wilcoxon signed rank test comparing the relative frequencies of responses on a 5-point Likert (distance, near) scale preferring AVA™ Smart program refraction and/or standard refraction assessment.
relative frequencies of scores | through study completion, an average of 8 weeks.
  P-value of Wilcoxon signed rank test comparing the relative frequencies of scores assessing lenses Essilor® AVA™ and non-AVA™ lenses following masked in-office trial (5-point Likert; Distance vision, Near work (phone reading), Computer, Across a room, Visual Comfort, Color Vision/Contrast Depth perception, Overall Quality of Vision, Overall satisfaction)
scores assessing lenses in Subjective Vision Quality | through study completion, an average of 8 weeks.
  P-value of Wilcoxon signed rank test comparing the relative frequencies of scores assessing lenses Essilor® AVA™/non AVA™ lenses in Subjective Vision Quality - OU (0-100 rating; Day driving, Night driving, Computer, across a room, Visual Comfort, Color Vision/Contrast, Depth Perception, Overall Quality of Vision, Adaptation speed, Ease of Adaptation, Overall satisfaction) following two weeks of wear.
scores assessing lenses evaluated by Patient (Preference) | through study completion, an average of 8 weeks.
  P-value of Wilcoxon signed rank test comparing the relative frequencies of scores assessing Essilor® AVA™/non-AVA™ lenses evaluated by Patient (Preference) - better confidence in refraction, higher satisfaction with refraction

CONTACTS AND LOCATIONS:
Overall Officials: Pete Kollbaum, Professor, Principal Investigator — Indiana University
Locations (1):
- Clinical Optics Research Lab @ Borish Center for Ophthalmic Research Indiana University School of Optometry Indiana University, Bloomington, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kollbaum PS, Jansen ME, Rickert ME. Comparison of patient-reported visual outcome methods to quantify the perceptual effects of defocus. Cont Lens Anterior Eye. 2012 Oct;35(5):213-21. doi: 10.1016/j.clae.2012.05.001. Epub 2012 May 28. PMID 22647932